CLINICAL TRIAL: NCT03603834
Title: Prospective Phase II Study of Neoadjuvant mFOLFOXIRI for Potentially Resectable Cholangiocarcinoma
Brief Title: Neoadjuvant mFOLFOXIRI for Potentially Resectable Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Jarin Chindaprasirt, Assistant professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE611336
Record Dates: First submitted 2018-07-17; First posted 2018-07-27 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cholangiocarcinoma
Keywords: Neoadjuvant; Potentially resectable; Chemotherapy; Bile duct cancer
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mFOLFOXIRI (Experimental): mFOLFOXIRI consists of the following combination of drugs:
  Oxaliplatin, 85 mg/m2, IV over 2 hours Leucovorin, 400 mg/m2, IV over 2 hours Irinotecan, 150 mg/m2, IV over 90 minutes 5 FU, 400 mg/m2, IV bolus 5FU, 2400 mg/m2, IV infusion over 46 hours after 5FU bolus injection
  each 14 day cycle, for 6 cycles
  Interventions: Drug: mFOLFOXIRI

INTERVENTIONS:
Drug: mFOLFOXIRI — mFOLFOXIRI consists of the following combination of drugs:
  1. Oxaliplatin, 85 mg/m2, IV over 2 hours
  2. Leucovorin, 400 mg/m2, IV over 2 hours
  3. Irinotecan, 150 mg/m2, IV over 90 minutes
  4. 5 FU, 400 mg/m2, IV bolus
  5. 5FU, 2400 mg/m2, IV infusion over 46 hours after 5FU bolus injection
  each 14 day cycle, for 6 cycles
  Other Names: Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

SUMMARY:
Previous reports suggest benefit of neoadjuvant chemotherapy/chemoradiation treatment for borderline resectable cholangiocarcinoma. This study is a single center prospective phase II study of neoadjuvant chemotherapy with mFOLFOXIRI in patients with borderline resectable cholangiocarcinoma.

DETAILED DESCRIPTION:
Previous reports suggest benefit of neoadjuvant chemotherapy/chemoradiation treatment for borderline resectable cholangiocarcinoma.

This study is a single center prospective phase II study of neoadjuvant chemotherapy with mFOLFOXIRI in patients with borderline resectable cholangiocarcinoma.

This phase 2 trial was designed to enroll 25 patients with BRCC who were assigned to mFOLFOXIRI neoadjuvant chemotherapy. The primary endpoint was the overall response rate.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Diagnosed with cholangiocarcinoma and the disease is measurable by RECIST 1.1 criteria
3. ECOG performance status of 0 or 1
4. No distant metastasis
5. The disease is either resectable or potentially resectable
6. Patients must have adequate organ function as defined by the following laboratory values at study entry:

   Hemoglobin ≥ 8 g/dL (transfusions are acceptable) ANC ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L AST/ALT ≤ 3 x ULN Total bilirubin ≤ 2.5 mg/dL Creatinine clearance ≥ 50 mL/min (estimated by Cockcroft-Gault or measured)
7. Women of childbearing potential definition (WOCBP) and men must agree to use adequate contraception prior, to study entry, for the duration of study participation, and 3 months after the end of treatment.
8. WOCBP must have a negative serum or urine pregnancy test prior to initiation of treatment.

Exclusion Criteria:

1. > 75 years old
2. Prior therapy for cholangiocarcinoma with either surgery, radiation or chemotherapy
3. Other malignancies except for the following: adequately treated cervical carcinoma in situ and treated basal cell carcinoma.
4. Hypersensitivity to 5FU, oxaliplatin (or other platinum agents), irinotecan (or to their excipients).
5. Pregnant or lactating women.
6. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
7. Liver disease including but not limited to cirrhosis, primary sclerosing cholangitis, future liver remnant of less than 20-30%
8. Comorbidity including but not limited to active clinically serious infections, congestive heart failure, life-threatening arrhythmia
9. known HIV positive
10. Baseline peripheral neuropathy/paresthesia grade ≥ 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The rate of overall response evaluated by MRI or CT | Up to 15 weeks
  The rate of response evaluated by MRI or CT according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Resectability rate | Up to 24 weeks
  The rate of patients who can successfully undergo surgery after chemotherapy
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | every 15 days for approximately 24 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jarin Chindaprasirt, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Jarin Chindaprasirt, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No